CLINICAL TRIAL: NCT03197350
Title: Characterization of Heart Failure With Preserved Ejection Fraction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HFpEF; 2012/23AVR/199 (Other: CEHF)
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure, Preserved Ejection Fraction; Cardiac Fibrosis; Biomarkers; Magnetic Resonance Imaging
Keywords: heart failure with preserved ejection fraction; Imaging; Prognosis
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — Biomarkers

STUDY DESIGN:
Intervention Model Description: The investigators will compare 3 different groups: controls and HFpEF patients and HFrEF patients, in order to better understand the pathophysiology in HF with preserved ejection fraction.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HFpEF (Active Comparator): We intend to recruit consecutive patients admitted for HFPEF in our institution during the next years. Eligible patients include those with age ≥50 years, LVEF ≥50%, symptomatic HF, and either a hospitalization for HF within the prior year or an elevated natriuretic peptide level (BNP ≥100 pg/mL or NT-proBNP ≥350 pg/mL) within the 60 days before inclusion.
  Intervention: cMR
  Interventions: Diagnostic Test: cMR; Biological: biomarker
- Controls (Active Comparator): We plan to recruit 10 per decade of age. These subjects will allow us to evaluate the effects of age on the parameters of our study. They will have no risk factors, a normal ECG at rest and normal heart ultrasound and no abnormalities on a stress test.
  Intervention: cMR
  Interventions: Diagnostic Test: cMR; Biological: biomarker
- HFrEF (Active Comparator): We intend to recruit consecutive patients admitted for HFrEF in our institution during the next years. Eligible patients include those with age ≥50 years, LVEF ≤40%, symptomatic HF, and either a hospitalization for HF within the prior year or an elevated natriuretic peptide level (BNP ≥100 pg/mL or NT-proBNP ≥350 pg/mL) within the 60 days before inclusion.
  Intervention: cMR
  Interventions: Diagnostic Test: cMR; Biological: biomarker

INTERVENTIONS:
Diagnostic Test: cMR — cardiac MRI done to complete the diagnosis
Biological: biomarker — Biomarker correlation with cMR parameters Prognostic information

SUMMARY:
The goals of this research will be to define some of the mechanisms underlying the progression and complications of heart failure (HF) with preserved left ventricular ejection fraction (HFPEF)

Aim 1: to evaluate the differences in cardiac structure, function and fibrosis markers through the spectrum of HF stages in order to deepen the understanding of the pathophysiology driving HF progression.

Aim 2: to define the mechanisms by which HF risk factors, such as hypertension, diabetes, obesity, and renal insufficiency, interact with age to increase HF risk, and to evaluate the role of precipitating factors such as myocardial ischemia, atrial fibrillation in HFPEF.

Aim 3: to determine prognostic factors in HFPEF patients, by following these patients over time. Accordingly the investigators will correlate baseline data (echocardiographic, MRI or biomarkers) with incident cardiovascular events and determine whether these measures provide incremental prognostic information beyond clinical characteristics.

DETAILED DESCRIPTION:
Heart failure (HF) is a prevalent and complex clinical syndrome characterized by significant morbidity and mortality. HF patients are classified into two major groups based on their left ventricular ejection fraction (LVEF): heart failure with reduced ejection fraction (HFrEF) (LVEF < 40%) and heart failure with preserved ejection fraction (HFpEF) (LVEF ≥ 50%). These groups exhibit distinct clinical and biological characteristics, and their underlying pathophysiology have been thoroughly investigated. However, HFpEF, which represents more than 50% of HF cases, remains a poorly understood disease with limited therapeutic options

Several proposed mechanisms contribute to the development of HFpEF, including systemic inflammation, microvascular dysfunction, cardiometabolic abnormalities, and interstitial fibrosis. The aim of our research programm is to understand the differences between the pathophysiology of this syndrome compared to that of heart failure with reduced EF, with a focus on cardiac fibrosis and metabolism.

ELIGIBILITY:
Controls without an history of HF and previous cardiovascular disease will be recruited

Inclusion Criteria for HF patients:

Patients need to have typical symptoms and signs of HF, New York Heart Association (NYHA) functional class II or higher, N-terminal pro-B type natriuretic peptide (NT-proBNP) >350pg/mL, or an hospitalization for HF within the previous 12 months. Left ventricular ejection fraction (LVEF) is required to be lower than 40% in patients with HFrEF and 50% or higher in HFpEF, with evident signs of diastolic dysfunction ( LA > 34 ml/m²; E/e' > 14; TR >2.8 ms, septal e' velocity < 7 cm/s or Lateral e' velocity <10 cm/s)

Exclusion Criteria for HF patients:

Patients with severe valvular disease, infiltrative or hypertrophic cardiomyopathy, acute coronary syndrome in the previous 30 days, chronic obstructive pulmonary disease GOLD 3 or 4, congenital heart disease, pericardial disease, terminal renal failure (eGFR < 15mL/min/1,73m²) or subjects requiring dialysis, atrial fibrillation with a ventricular response > 140 bpm, severe anemia (hemoglobin < 8 g/dL), liver dysfunction, and evolving cancer will be excluded

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-12-04 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Prognosis with a follow up including HF hospitalizations and/or deaths. | 6 months
  A follow up will be done by the investigators. After that, they will determine if fibrosis estimated by cMR or biomarkers is a significant prognostic factor.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Catherine Pouleur, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint Luc, Brussels, Belgium

REFERENCES:
- [Derived] de Terwangne C, Menghoum N, Boute M, Lejeune S, Pasquet A, Gerber B, Vancraeynest D, Boland B, Beauloye C, Pouleur AC. Heart failure with preserved ejection fraction shows no excess mortality in older patients: a population-matched relative survival analysis. Geroscience. 2026 Jan 6. doi: 10.1007/s11357-025-02063-0. Online ahead of print. PMID 41495328
- [Derived] Menghoum N, Badii MC, Leroy M, Parra M, Roy C, Lejeune S, Vancraeynest D, Pasquet A, Brito D, Casadei B, Depoix C, Filippatos G, Gruson D, Edelmann F, Ferreira VM, Lhommel R, Mahmod M, Neubauer S, Persu A, Piechnik S, Hellenkamp K, Ikonomidis I, Krakowiak B, Pieske B, Pieske-Kraigher E, Pinto F, Ponikowski P, Senni M, Trochu JN, Van Overstraeten N, Wachter R, Gerber BL, Balligand JL, Beauloye C, Pouleur AC. Exploring the impact of metabolic comorbidities on epicardial adipose tissue in heart failure with preserved ejection fraction. Cardiovasc Diabetol. 2025 Mar 22;24(1):134. doi: 10.1186/s12933-025-02688-7. PMID 40121452
- [Derived] Lejeune S, Ginion A, Menghoum N, Vancraeynest D, Pasquet A, Gerber BL, Horman S, Beauloye C, Pouleur AC. Association of Plasma Myeloperoxidase with Inflammation and Diabetic status in HFpEF. Rev Cardiovasc Med. 2023 Feb 8;24(2):56. doi: 10.31083/j.rcm2402056. eCollection 2023 Feb. PMID 39077419
- [Derived] Roy C, Slimani A, de Meester C, Amzulescu M, Pasquet A, Vancraeynest D, Beauloye C, Vanoverschelde JL, Gerber BL, Pouleur AC. Associations and prognostic significance of diffuse myocardial fibrosis by cardiovascular magnetic resonance in heart failure with preserved ejection fraction. J Cardiovasc Magn Reson. 2018 Aug 8;20(1):55. doi: 10.1186/s12968-018-0477-4. PMID 30086783